CLINICAL TRIAL: NCT00342264
Title: Diesel Exhaust in Miners Study
Brief Title: A Nested Case-Control Study of Lung Cancer and Diesel Exhaust Among Non-Metal Miners
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999003; OH99-C-N003
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Occupational Cohort; Diesel Exhaust; Natural History
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: The study cohort will be comprised of underground, and surface workers (excluding administrative workers) who have been employed in the candidate non-metal mines for at least one year during the period between the date of dieselization of each mine and December 31, 1996.

SUMMARY:
Diesel exhaust has been classified as a probable carcinogen by the International Agency for Research on Cancer and as a potential carcinogen by the National Institute for Occupational Safety and Health (NIOSH). The carcinogenicity of this pollutant is of concern not only for the one million workers who are exposed occupationally, but also for the general population. Over 30 epidemiologic studies of diesel exhaust exposure have been performed, and the results suggest an increase in lung cancer risk. However, the association is not well defined. Past studies have suffered from the use of crude indicators of exposure, inadequate control of confounding, and/or short follow-up periods, low exposure levels, and small numbers of observations.

NCI and NIOSH are collaborating on two related studies of diesel exhaust under the NCI/NIOSH Interagency Agreement. First, a retrospective cohort mortality study of about 8,200 non-metal miners will be performed to investigate lung cancer mortality in relation to quantitative measures of diesel exhaust exposure, and to determine whether there is evidence of elevated mortality from other causes of death among diesel exhaust exposed miners. The retrospective cohort study will be performed using existing records and information and has been exempted from IRB review. NIOSH is the lead agency on the retrospective cohort study.

The proposed study is a case-control study nested in the retrospective cohort of non-metal miners. The study is expected to include at least 160 members of the cohort who died from lung cancer and four matched controls for each case. Using a structured questionnaire, detailed information will be collected on each subject's lifetime exposure to diesel exhaust, as well as information on smoking and other confounders. This information will allow investigators to examine the association between lung cancer and different quantitative measures of diesel exhaust exposure, adjusted for smoking and other potential confounders.

DETAILED DESCRIPTION:
Diesel exhaust has been classified as a probable carcinogen by the International Agency for Research on Cancer and as a potential carcinogen by the National Institute for Occupational Safety and Health (NIOSH). The carcinogenicity of this pollutant is of concern not only for the one million workers who are exposed occupationally, but also for the general population. Over 30 epidemiologic studies of diesel exhaust exposure have been performed, and the results suggest an increase in lung cancer risk. However, the association is not well defined. Past studies have suffered from the use of crude indicators of exposure, inadequate control of confounding, and/or short follow-up periods, low exposure levels, and small numbers of observations.

NCI and NIOSH are collaborating on two related studies of diesel exhaust under the NCI/NIOSH Interagency Agreement. First, a retrospective cohort mortality study of about 8,200 non-metal miners will be performed to investigate lung cancer mortality in relation to quantitative measures of diesel exhaust exposure, and to determine whether there is evidence of elevated mortality from other causes of death among diesel exhaust exposed miners. The retrospective cohort study will be performed using existing records and information and has been exempted from IRB review. NIOSH is the lead agency on the retrospective cohort study.

The proposed study is a case-control study nested in the retrospective cohort of non-metal miners. The study is expected to include at least 160 members of the cohort who died from lung cancer and four matched controls for each case. Using a structured questionnaire, detailed information will be collected on each subject's lifetime exposure to diesel exhaust, as well as information on smoking and other confounders. This information will allow investigators to examine the association between lung cancer and different quantitative measures of diesel exhaust exposure, adjusted for smoking and other potential confounders.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Subjects will be identified from all 10 mines participating in the cohort study.

Cases from each mine will be lung cancer deaths as specified on the death certificate occurring among members of the cohort working at the mine between the date the mine was dieselized and December 31, 1996.

Children will be excluded from participating.

We will exclude cases that are found either not likely to be carcinoma of the lung or metastatic to the lung by slide review or pathology report.

Four controls will be selected for each case by random sampling from among all members of the cohort who were alive prior to the day the case died.

Controls will be individually matched to the case on mine, gender, race/ethnicity, and year of birth (within 5 years).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Diesel Exhaust in Miners Study (DEMS) is a cohort study of 12,315 nonmetal miners employed in 8 study mines (3 trona mines in Wyoming, 3 potash mines in New Mexico, 1 limestone mine in Missouri and 1 salt mine in Ohio), coupled with a nested case-control study of lung cancer to obtain information on smoking and other potential confounders from telephone interviews with next of kin of all cases and dead controls and direct interviews with living controls.
Sampling Method: Non-Probability Sample
Enrollment: 1187 (Actual)
Dates: Start 1999-01-12 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Lung cancer death | death
  Lung cancer death

CONTACTS AND LOCATIONS:
Overall Officials: Debra Silverman, D.Sc., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Westat Inc, Rockville, Maryland, United States